CLINICAL TRIAL: NCT06718855
Title: Cognitive Functioning in People with Myasthenia Graivs: Impact on Daily Life Activities, Work, Disability and Quality of Life
Acronym: MYCOG
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: MYCOG
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Cognitive Functioning; Disability; Activities of Daily Living; Quality of Life; Anxiety; Comorbidities; Work; Depression; Memory; Attention; Executive Functions; Cognitive Reserve
MeSH Terms: conditions — Myasthenia Gravis; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
MYCOG primarily aims to estimate the prevalence of cognitive difficulties in patients with MG treated at Besta Institute. Secondary aims include: a) assess the degree to which cognitive difficulties are associated to work impairment, limitations in ADL, symptoms of anxiety and depression, fatigue, disability and QoL; b) assess whether patients with different MG types show different degrees of cognitive impairment; c) assess whether patients with different MG antibody profiles show different degrees of cognitive impairment; d) assess whether patients under different MG-specific pharmacological treatments show different degrees of cognitive impairment.

DETAILED DESCRIPTION:
Previous literature findings provide contradictory indications about presence of cognitive impairment in patients with MG, but patients experience different degree of limitations in ADLs, disability and QoL which might not be entirely understood on the basis of neuromuscular symptoms. We therefore aimed to address the potential impact of cognitive impairment.

MYCOG is a monocentric, cross-sectional and observational study which primarily aims to estimate the prevalence of cognitive difficulties, measured with Global Examination of Mental State (GEMS), in patients with MG treated at Besta Institute. Secondary aims include: a) assess the degree to which cognitive difficulties are associated to work impairment (measured with WPAI-GH), limitations in ADL (measured with MG-ADL), symptoms of anxiety and depression (measured with HADS), fatigue (measured with FSS), disability and QoL (measured with MG-DIS and MG-QOL15); b) assess whether patients with different MG types (ocular, generalized, bulbar, pharmacological remission and clinical stable remission) show different degrees of cognitive impairment; c) assess whether patients with different MG antibody profiles (AChR, MuSK, Double Negative) show different degrees of cognitive impairment; d) assess whether patients under different MG-specific pharmacological treatments (piridogstigmine, steroids, other therapies such as immunemodulators) show different degrees of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MG,
* followed-up at Besta institute
* aged 18-99,
* able to understand Italian language;

Exclusion Criteria:

* psychiatric comorbidies of psychotic nature;
* do not accept to participate on a voluntary basis;
* patients who should be excluded based on physician's judgement;
* patients who live in a nursing home for aged or disabled persons;
* respiratory impairment (patients under mechanical ventilation)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Italian speakers, already followed at Besta Institute
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
GEMS | 22 months
  Global examination of cognitive functioning

SECONDARY OUTCOMES:
CRIq | 22 months
  Cognitive reserve index
ENB-3 | 22 months
  Brief Neuropsychological battery
MG-DIS | 22 months
  Disability
MG-QOL15 | 22 months
  Quality of life
MG-ADL | 22 months
  Activities of Daily Living
WPAI-GH | 22 months
  Impact on work-related activities and productivity
HADS | 22 months
  Anxiety and depression
FSS | 22 months
  Fatigue Severity
CCI | 22 months
  Presence of comorbidities
Clinical profile | 22 months
  General information on MG type, antibody profile, sociodemographic information, MG-specific symptoms, pharmacological therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No